CLINICAL TRIAL: NCT02898168
Title: The Therapeutic Effects of Peroneal Nerve Functional Electrical Stimulation for Lower Extremity in Patients With Sub-acute Post-stroke Hemiplegia A Randomized Controlled Study
Brief Title: The Therapeutic Effects of Peroneal Nerve Functional Electrical Stimulation for Lower Extremity in Patients With Sub-acute Post-stroke Hemiplegia
Acronym: RALLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Nippon Medical School (Other); Kagoshima University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIORTHO1524; UMIN-CTR (Other: UMIN000020604)
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: stroke; Rehabilitation; WalkAide (WA); Functional Electrical Stimulation (FES)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WA (Experimental)
  Interventions: Device: WA group
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Device: WA group — Conventional rehabilitation therapy and gait training with WAIntervention with WA is scheduled 40min/day, five times a week, for 8 weeks.
  Arms: WA
Other: Control — Conventional rehabilitation therapy and gait training without WA.
  Arms: Control

SUMMARY:
Among the sequelae of stroke, gait disorder is directly linked to the degree of autonomy in the daily life of patients. It is considered significant effects on their Quality of Life(QOL).

Further methods of rehabilitation are required for convalescent patients to recover their function soon and better, due to a multitudes of recovery patient with troubles such as gait problem.

This trial is studying to investigate the effects of gait training with a functional electrical stimulation (FES) 'WalkAide[R](WA)' to improve the lower-limb function and ambulation in convalescent stroke patients.

DETAILED DESCRIPTION:
This study is targeting convalescent patients within 6 months after the onset of initial stroke (cerebral infarction or cerebral hemorrhage) and also observing the foot drop during walking.

Some study for the patients after the onset of stroke (over several months) are reported that a case of the efficacy by the treatment using the FES, and another case of using FES indicated the equal efficacy and the higher QOL compared to using ankle-foot orthosis(AFO).

However, these are clinical research results overseas and there are not so many studies targeting only for convalescent stroke patients.

FES which recover the lost function by paralysis using electrical stimulation is recommended as convalescent rehabilitation by Japanese Guidelines for the Management of Stroke 2015 etc..

The purpose of FES treatment is the electrical stimulation to peroneal nerve of patients with foot drop and equinus foot due to central nervous system damage and the objective efficacy is following:

* To improve the walking by dorsiflexing the foot during swing phase
* To prevention and suppression of disuse atrophy
* To increase local blood flow
* To re-educate muscle
* To maintain or increase the range of joint motion

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients who agree to participate in this study and provide their informed consent
* 2) Patients from 20 to 85 years old at the time of consent
* 3) Patients of convalescent stoke (within 6 months of onset)
* 4) Patients with a first episode of stroke, which type limited intracranial hemorrhage or ischemic stroke (excluding subarachnoid hemorrhage)
* 5) Patients inpatients for the rehabilitation therapy
* 6) Patients diagnosed 3 or 4 on Functional Ambulation Classification (FAC)
* 7) Patients stable general condition(blood pressure, pulse, blood glucose level etc.)
* 8) Patients with drop foot in walking

Exclusion Criteria:

* 1) Patients due to severe heart disease
* 2) Patients with previous gait disability, such as neurological disease
* 3) Patients with previous orthopedic disease, such as knee osteoarthritis
* 4) Patients with severe hepatic or renal dysfunction
* 5) Patients with severe sensory disturbance or severe ataxia or severe higher brain dysfunction
* 6) Patients correspond to contraindicated for the electrical stimulation (e.g. patients with a medical implant or implantable medical electrical equipment such as a cardiac pacemaker)
* 7) Patients with severe skin disease
* 8) Patients with any dose adjustment of antispasticity drugs (tizanidine hydrochloride, eperisone hydrochloride, baclofen, etc.) within 1month
* 9) Patients whose impairment severities changed during the study period
* 10) Patients taking the botulinum toxin formulation injection or the nerve block injection with phenol within 6months
* 11) Patients with any lower limb treatment using FES or the robot suit within 1month
* 12) Patients diagnosed not to use during the the WA trial operation period
* 13) Patients who do not complete the WA trial operation for 7 days
* 14) Patients joining any other clinical trials or studies with intervention

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
maximum walking distance of 6 Minute Walk Test (bare feet) | 8weeks
  Measuring maximum walking distance of 6 Minute Walk Test at baseline and after 8-weeks intervention. Calculating difference of those measured values. Targeting for all patients.

SECONDARY OUTCOMES:
maximum walking distance of 6 Minute Walk Test (with WA) | 8weeks
  Measuring maximum walking distance of 6 Minute Walk Test at baseline and after 8-weeks intervention. Calculating difference of those measured values.
  Targeting only for WA group.
maximum walking distance of 6 Minute Walk Test (with AFO) | 8weeks
  Measuring maximum walking distance of 6 Minute Walk Test at baseline and after 8-weeks intervention. Calculating difference of those measured values.
  Targeting only for patients using AFO before starting this study.
walking speed of 10 Meter Walk Test (bare feet) | 8weeks
  Measuring maximum walking speed of 10 Meter Walk Test at baseline and after 8-weeks intervention. Calculating difference of those measured values. Targeting for all patients.
walking speed of 10 Meter Walk Test (with WA) | 8weeks
  Measuring maximum walking speed of 10 Meter Walk Test at baseline and after 8-weeks intervention. Calculating difference of those measured values. Targeting only for WA group.
walking speed of 10 Meter Walk Test (with AFO) | 8weeks
  Measuring maximum walking speed of 10 Meter Walk Test at baseline and after 8-weeks intervention. Calculating difference of those measured values. Targeting only for patients using AFO before starting this study.
Fugl-Meyer assessment (FMA) | 8weeks
  Calculating difference of the total score of lower extremity subscale of the Fugl-Meyer Assessment (perfect score: 34 points) at baseline and after 8-weeks intervention.
modified Ashworth scale (MAS) | 8weeks
  Calculating difference of the muscle tone six levels ( 0 , 1 , 1+ , 2 , 3 , 4 ) at baseline and after 8-weeks intervention.
range of motion | 8weeks
  Calculating difference of the angle of the ankle succumbed back (5 ° increments) at baseline and after 8-weeks intervention.
Timed up and go test (bere feet) | 8weeks
  Measuring the time that patients take to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down .
  Calculating difference of those measured values between at baseline and after 8-weeks intervention. Targeting for all patients.
Timed up and go test (with AFO) | 8weeks
  Measuring the time that patients take to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down .
  Calculating difference of those measured values between at baseline and after 8-weeks intervention. Targeting only for patients using AFO before starting this study.
Timed up and go test (with WA) | 8weeks
  Measuring the time that patients take to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down .
  Calculating difference of those measured values between at baseline and after 8-weeks intervention. Targeting only for WA group.
Stroke Impact Scale (SIS) | 8weeks
  An evaluation of summation score of the total score and physical domain (sixth domain) score. Calculating difference of those measured values between at baseline and after 8-weeks intervention.
Patient reported outcome measure (PRO) | 8weeks
  Evaluation gait analysis using visual analogue scale(VAS scale) by Patient's own. Calculating the difference of these VAS scale between at baseline and after 8-weeks intervention.
gait analysis by medical staff | 8weeks
  Evaluation using total score of gait analysis by medical staff (-48~48).Calculating difference of these score between at baseline and after 8-weeks intervention.
Adverse event assessment | 8weeks
  A frequency counting of the adverse events. LLT code will be assigned to the reported adverse event using the MedDRA dictionary.
  The origin date of the term until adverse events define the start date of the treatment program(0 week).
  Also doing a frequency counting of adverse events observed during the the WA trial operation period, but not included in the safety evaluation of the treatment program.

CONTACTS AND LOCATIONS:
Overall Officials: Shuji Matsumoto, MD, Ph.D, Study Chair — Nippon Medical School
Locations (31):
- Japan (31):
  - Shinyachiyo Hospital, Yachiyo, Chiba
  - Matsuyama Rehabilitation Hospital, Matsuyama, Ehime
  - St.Mary's Hospital Healthcare Center, Kurume, Fukuoka
  - Yame Rehabilitation Hospital, Yame, Fukuoka
  - Hokusei Memorial Hospital, Kitami, Hokkaido-prefecture
  - Ohkawara Neurosurgical Hospital, Muroran, Hokkaido-prefecture
  - Tokachi Rehabilitation Center, Obihiro, Hokkaido-prefecture
  - Sapporo Shiroishi Memorial Hospital, Sapporo, Hokkaido-prefecture
  - Sapporo Keijinkai Rehabilitation Hospital, Sapporo, Hokkaido-prefecture
  - Tokeidai Memorial Hospital, Sapporo, Hokkaido-prefecture
  - Yoshida Hospital, Cerebrovascular Research Institute, Kobe, Hyōgo
  - Kajikionsen Hospital, Aira, Kagoshima-ken
  - Acras Central Hospital, Kagoshima, Kagoshima-ken
  - Department of Rehabilitation and Physical Medicine, Graduate School of Medical and Dental Sciences, Kagoshima University, Kagoshima, Kagoshima-ken
  - Kohshinkai Ogura Hospital, Kanoya, Kagoshima-ken
  - Tarumi City Medical Center Tarumi Central Hospital, Tarumizu, Kagoshima-ken
  - Sakura Jyuji Hospital, Kumamoto, Kumamoto
  - Kumamoto Takumadai Rehabilitation Hospital, Kumamoto, Kumamoto
  - Fujimotokanmachi Hospital, Miyakonojō, Miyazaki
  - Junwakai Memorial Hospital, Miyazaki, Miyazaki
  - Nichinan Municipal Chubu Hospital, Nichinan, Miyazaki
  - Yohkoh Rehabilitation Hospital, Sasebo, Nagasaki
  - Nagasakikita Hospital, Togitsu-cho, Nishisonogi-gun, Nagasaki
  - Chuzan Hospital, Okinawa, Okinawa
  - Okinawa Rehabilitation Center Hospital, Okinawa, Okinawa
  - Nanbu-Tokushukai Hospital, Shimajiri-gun, Okinawa
  - Kansai Rehabilitation Hospital, Toyonaka, Osaka
  - Saitama Misato Sogo Rehabilitation Hospital, Misato, Saitama, Saitama
  - Seirei Hamamatsu City Rehabilitaion Hospital, Hamamatsu, Shizuoka
  - Hakujikai Memorial Hospital, Adachi-ku, Tokyo
  - IMS Itabashi Rehabilitation Hospital, Itabashi-ku, Tokyo